CLINICAL TRIAL: NCT00818727
Title: Bone Density of Newborn Infants to Mothers Treated With Selective Serotonin Reuptake Inhibitor (SSRI)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr.Ayala Maayan, sheba medical center
Other Study IDs: SHEBA-09-5435-AM-CTIL
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Last update posted 2009-01-08 (Estimated); Status verified 2009-01

CONDITIONS: Bone Density
Keywords: Bone density; SSRI; newborn infants

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
SSRI treatment in adults was found to decrease bone density. The use of SSRI among pregnant women with depression or anxiety is extendent and raising. The effect of bone density of the infants was not yet evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Term newborn infants to mothers treated with SSRI and healthy controls

Exclusion Criteria:

* Preterms, major congenital malformations.

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Healthy term newborn infants to mothers treated with SSRI and healthy controls. bone density mesurment will be applied on the 1-7 days of life.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
bone density | 1 month
bone density | 2 years